CLINICAL TRIAL: NCT05410379
Title: Antral Lesions Characterization of a New Cryoballoon Ablation System in Terms of Local Impedance Drop
Acronym: CryoLID
Status: Completed | Type: Observational
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MCH 2021-01
Record Dates: First submitted 2022-06-01; First posted 2022-06-08 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial fibrillation (AF) is defined as a supraventricular tachyarrhythmia with uncoordinated atrial electrical activation and consequently ineffective atrial contraction. Electrocardiographic characteristics of AF include: irregularly irregular R-R intervals (when atrioventricular conduction is not impaired), absence of distinct repeating P waves, and irregular atrial activations.

Different AF classifications have been proposed but, traditionally, four patterns of AF are distinguished, based on presentation, duration, and spontaneous termination of AF episodes. Paroxysmal AF, that terminates spontaneously or with intervention within 7 days of onset. Persistent AF that is continuously sustained beyond 7 days, including episodes terminated by cardioversion (drugs or electrical cardioversion) after >7 days. Long-standing persistent (continuous AF of >12 months' duration) when decided to adopt a rhythm control strategy. Permanent AF, that is accepted by the patient and physician, and no further attempts to restore/maintain sinus rhythm will be undertaken.

The purpose of this study is to perform assessments of local impedance before and after cryoablation performed with the new POLAR X cryoballoon, in order to characterize the quality of the lesion and possibly to associate it with the acute success and 12 months AF recurrence-free rate.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects indicated for the treatment of AF with the cryoablation system according to current and future Guidelines and system indications for use;
2. Subjects who are willing and capable of providing informed consent;
3. Subjects who are willing and capable of participating in all testing associated with this clinical study at an approved clinical investigational center.
4. Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Any known contraindication to an AF ablation or anticoagulation, including those listed in the instructions for use;
2. Subjects with indication for treatment of AF that is not according to current and future Guidelines and system indications for use;
3. Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause;
4. Known or pre-existing severe Pulmonary Vein Stenosis;
5. Evidence of myxoma, LA ( left atrium) thrombus or intracardiac mural thrombus;
6. Previous cardiac surgery (e.g. ventriculotomy or atriotomy, CABG (Coronary artery bypass graft surgery ), PTCA ( Percutaneous transluminal coronary angioplasty), stent procedure) within 90 days prior to enrollment;
7. Implantable cardiac device procedures ,e.g. PM (pacemaker), ICD( implantable cardioverter defibrillators), CRT within 30 days prior to enrollment;
8. Implanted Left Atrial Appendage Closure device prior to the index procedure;
9. Interatrial baffle, closure device, patch, or patent foramen ovale (PFO) occluder;
10. Subjects with severe valvular disease OR with a prosthetic - mechanical or biological

    - heart valve (not including valve repair and annular rings);
11. Presence of any pulmonary vein stents;
12. Active systemic infection;
13. Vena cava embolic protection filter devices and/ or known femoral thrombus;
14. Any previous history of cryoglobulinemia;
15. History of blood clotting or bleeding disease;
16. Any prior history of documented cerebral infarct, TIA (transient ischemic attack) or systemic embolism (excluding a post-operative deep vein thrombosis (DVT)) ≤ 180 days prior to enrollment;
17. Subjects who are hemodynamically unstable or with structural heart disease;
18. The subject is unable or not willing to complete follow-up visits and examination for the duration of the study;
19. Life expectancy ≤ 1 year per investigator's opinion;
20. Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon investigator's discretion);
21. Unrecovered/unresolved Adverse Events from any previous invasive Procedure;
22. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in the CryoLID study will be clinically indicated for a cryoablation procedure and meet the study inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
local impedance drop | 6 months
  The primary endpoint of the study is the local impedance drop, measured as the difference between local impedance recorded by the rhythmic HDx mapping system at baseline and after PVI (pulmonary vein isolation) . For the primary endpoint assessment, impedance data will be analyzed offline and grouped per 4 anatomical segments around each pulmonary vein (PV). Absolute values of local impedance measured at baseline and after PVI, as well as local impedance drops will be also compared according to lesion success and according to the value of conventional predictors of successful cryo-lesions (e.g. TTI ( time to isolation ) < 60 s).

SECONDARY OUTCOMES:
failure-free rate at 12 months | 12 months.
  The endpoint is the recurrence of atrial tachycardia (AT) and AF after the blanking period (3 months), as measured by means of ECG and 24h-holter. It will be evaluated by the failure-free rate at 12 months post-index procedure in each cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- MCH, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No